CLINICAL TRIAL: NCT01492387
Title: Individualizing Duration of Antibiotic Therapy in Hospitalized Patients With Community - Acquired Pneumonia: a Non-inferiority, Randomized, Controlled Trial.
Brief Title: Duration of Antibiotic Therapy in Community - Acquired Pneumonia
Acronym: DURATION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Francesco Blasi, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DURATION
Record Dates: First submitted 2011-12-05; First posted 2011-12-15 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Pneumonia; Bronchopneumonia; Pleuropneumonia; Pneumonia, Bacterial; Pneumonia, Viral
Keywords: community-acquired pneumonia; healthcare-associated pneumonia; antibiotic therapy; Duration of therapy
MeSH Terms: conditions — Pneumonia; Bronchopneumonia; Pleuropneumonia; Pneumonia, Bacterial; Pneumonia, Viral; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local standard of care (No Intervention): Patients randomized to this arm will be treated for the duration of therapy dictated by the primary care physician.
- Individualized arm (Experimental): Patients randomized to this arm will be treated according to clinical response: antibiotic therapy will be discontinued 48 hours after the day that the patient reaches clinical stability, with at least 5 days of total antibiotic treatment.
  Interventions: Other: Discontinuation of antibiotic therapy

INTERVENTIONS:
Other: Discontinuation of antibiotic therapy — Patients randomized in the Individualized Arm will be treated according to clinical response: antibiotic therapy will be discontinued 48 hours after the day that the patient reaches clinical stability, with at least 5 days of total antibiotic treatment.
  Arms: Individualized arm

SUMMARY:
The purpose of the study is to assess the efficacy of an individualized approach to duration of antibiotic therapy based on each subject's clinical response compared to a local standard approach in patients coming from the community and who are hospitalized because of a pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Patients will be 18 years old or older and meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Diagnosis of pneumonia:

   Evidence of a new pulmonary infiltrate seen on either radiograph or computed tomography of the chest within 48 hours after hospitalization plus at least two among the following: 1) new or increased cough with/without sputum production and/or purulent respiratory secretions; 2) fever (documented temperature -rectal or oral- ≥ 37.8 °C) or hypothermia (documented temperature -rectal or oral- <36o C); 3) deterioration of oxygenation; 4) evidence of systemic inflammation (such as abnormal white blood cell count -either leukocytosis (>10,000/cm3) or leukopenia (< 4,000/cm3) - or increasing of C-reactive protein or procalcitonin values above the local upper limit.

   CAP will be defined as pneumonia occurring in any patient admitted to the hospital coming from the community and who were not hospitalized in the previous 14 days. HCAP will be defined as a community-acquired pneumonia occurring in a patient with any of the following special epidemiological characteristics: patient who was hospitalized for 2 days or more in the previous 90 days; patient coming from a nursing home or extended care facility; patient who received home infusion therapy (including antibiotics) or wound care in the previous 30 days; patient who was on chronic dialysis in the previous 30 days.
2. An appropriate empiric antibiotic therapy for the pneumonia received within 24 hours after admission to the hospital.
3. A clinical stability reached within 5 days after hospital admission, in the absence of any changes of the initial empiric antibiotic therapy.
4. Signed informed consent

Exclusion Criteria:

Patients presenting with any of the following will not be included in the trial:

1. Patients with immunodeficiency, defined as: chemotherapy in the previous 12 months, radiotherapy in the previous 12 months, transplantation, immunosuppressive treatment, hematologic malignancy, AIDS or HIV with CD4 count < 200, asplenia.
2. Patients with a concomitant infection on admission to the hospital requiring antibiotic therapy (i.e urinary tract infection). The presence of sepsis due to pneumonia will not be considered another concomitant infection.
3. Patients with documented bacteremia due to S. aureus in a blood culture (both methicillin resistant and susceptible S. aureus)
4. Patients with etiology of pneumonia due to fungi, mycobacterium or Pneumocystis jiroveci.
5. Patients hospitalized in the previous 15 days

Inclusion and exclusion criteria for the proposed study will not limit the study cohort on the basis of sex, ethnicity, socioeconomic status or other potentially discriminatory factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Composite outcome including adverse events | 30 days
  Any among the following: 1) disease-specific complications due to pneumonia, such as lung abscess, empyema, meningitis, endocarditis, arthritis or pericarditis; 2) clinical failure during hospitalization (either hemodynamic or respiratory failure); 3) a new course of antibiotics (at least one dose), after discontinuation of antibiotic therapy given for the pneumonia, either endovenous or oral; 4) re-hospitalization; 5) death.

SECONDARY OUTCOMES:
Composite outcome of other adverse events | 30 days
  Any among the following: 1) disease-specific complications due to pneumonia, such as lung abscess, empyema, meningitis, endocarditis, arthritis or pericarditis; 2) clinical failure due to pneumonia occurring during hospitalization (either hemodynamic or respiratory failure); 3) a new course of antibiotics (at least one dose), after discontinuation of antibiotic therapy given for the pneumonia, either endovenous or oral, for a relapse of pneumonia; 4) re-hospitalization due to a relapse of pneumonia; 5) death due to pneumonia.
Antibiotic exposure | 90 days
  Days of antibiotic exposure, including intravenous and oral antibiotic therapy given for any reason.
Adverse effects | 90 days
  Adverse effects will include: anaphylactic reactions and allergic skin reactions; Clostridium difficile-associated colitis; hematologic toxicity; hepatotoxicity; convulsions; tendinopathies; peripheral neuropathy; prolongation of the QTc interval; nausea; diarrhea; vomiting; abdominal pain; nephrotoxicity.
Composite outcome of other adverse events at 90 days | 90 days
  Any among the following: 1) a new course of antibiotics for any reason after discontinuation of antibiotic therapy for pneumonia; 2) re-hospitalization for any reason; 3) death from any reason.
Length of hospitalization | 30 days
  Number of days from the date of admission to the hospital to either the date of discharge (patients sent home or to a long-term care facility) or the date of death if occurred during hospitalization.
Costs | 30 days
  Costs of care differences between the two study groups based on the total length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Aliberti, MD, Principal Investigator — University of Milano Bicocca, Milan, Italy; Julio A Ramirez, MD, Principal Investigator — University of Louisville, KY, USA
Locations (15):
- Italy (15):
  - AO Ospedali Riuniti Bergamo, Bergamo
  - AO Policlinico S. Orsola Malpighi, University of Bologna, Bologna
  - AO S. Anna, Como
  - University of Genoa, Genoa
  - AO C. Poma, Mantova
  - AO San Carlo Borromeo, Milan
  - IRCCS Fondazione Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Luigi Sacco, University of Milan, Milan
  - University of Modena e Reggio Emilia, Modena
  - Univeristy of Milano Bicocca, Monza
  - IRCCS Policlinico S. Matteo, University of Pavia, Pavia
  - AO S. Maria Nuova, Reggio Emilia
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico di San Donato Milanese, University of Milan, San Donato Milanese
  - AO S. Maria della Misericordia,, Udine

REFERENCES:
- [Background] Aliberti S, Blasi F, Zanaboni AM, Peyrani P, Tarsia P, Gaito S, Ramirez JA. Duration of antibiotic therapy in hospitalised patients with community-acquired pneumonia. Eur Respir J. 2010 Jul;36(1):128-34. doi: 10.1183/09031936.00130909. Epub 2009 Nov 19. PMID 19926738
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Woodhead M, Blasi F, Ewig S, Garau J, Huchon G, Ieven M, Ortqvist A, Schaberg T, Torres A, van der Heijden G, Read R, Verheij TJ; Joint Taskforce of the European Respiratory Society and European Society for Clinical Microbiology and Infectious Diseases. Guidelines for the management of adult lower respiratory tract infections--full version. Clin Microbiol Infect. 2011 Nov;17 Suppl 6(Suppl 6):E1-59. doi: 10.1111/j.1469-0691.2011.03672.x. PMID 21951385